CLINICAL TRIAL: NCT06697574
Title: HypnOLP Trial Hypnotherapy for Oral Lichen Planus - a Single Blind Randomized Controlled Trial
Brief Title: Hypnotherapy for Oral Lichen Planus. Patients with Clinically and Histologically Confirmed Oral Lichen Planus Would Be Randomized for Hypnotherapy Vs Psychoeducation About the Pyschoneuroimmune System. Follow Up Would Be Done At 2, 6, 12 Weeks After.
Acronym: HypnOLP
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TASMC-24-GW-0299-CTIL
Record Dates: First submitted 2024-11-11; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Oral Lichen Planus
Keywords: Oral Lichen Planus; Hypnosis
MeSH Terms: conditions — Lichen Planus, Oral

STUDY DESIGN:
Intervention Model Description: 60 randomised patients as well as 30 retrospective
Who Masked: Care Provider
Masking Description: Original care providers who are preforming the follow up would be blinded to the intervention. The provider of the intervention is not aware of the state of the lichen planus of each patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Psychoeducation and Hypnotherapy Group (Experimental): 30 Patients randomized to undergo psychoeducation and hypnotherapy
  Interventions: Behavioral: Hypnosis aimed at stress reduction and health of the oral mucosa; Behavioral: Psychoeducation
- Psychoeducation Group (Active Comparator): 30 Patients selected for psychoeducation with out hypnotherapy
  Interventions: Behavioral: Psychoeducation
- Non intervention group - retrospectively analyzed (No Intervention): 30 age matched patients from the oral mucosal clinic who's course and presentation of lichen planus would be retrospectively analyzed

INTERVENTIONS:
Behavioral: Hypnosis aimed at stress reduction and health of the oral mucosa — * Induction.
  * Hypnotic relaxation and escalating deepening of hypnotic trance.
  * Suggestions for healing and wellness of the oral mucosa and for balanced and optimal performance of the immune system, tailoring metaphors and images based on interview with patients.
  "…the interior of the mouth is soft, healthy pink, intact and whole. It functions optimally as it should - enabling joyful eating and tasting, speaking with ease for any needed expression, any function of the mouth that needs to be used can be done so easily.
  The immune system is very wise - it knows perfectly how to function in a balanced and harmonious way. Its wisdom enables it to act if the body needs defense and to standby and rest if it does not".
  * Ego strengthening.
  * Anchoring - using a predetermined mark selected by the patient.
  * Dehypnotisation.
  Arms: Psychoeducation and Hypnotherapy Group
Behavioral: Psychoeducation — A short explanation about the psycho-neuro-immune system and its part in oral lichen planus
  Arms: Psychoeducation Group; Psychoeducation and Hypnotherapy Group

SUMMARY:
60 patients with clinically and histologically confirmed Oral Lichen Planus, which are are typically followed up at our oral mucosal disease clinic with a standing diagnosis for at least 1 year would be randomized.

30 would undergo a session of psychoeducation and hyponotherapy and 30 would undergo psychoeducation alone. This would be done by the PI who is an oral medicine specialist and licensed for medical hypnosis.

Patients would be instructed to practice self hypnosis and would be followed up by their original oral medicine specialists who would be blinded to the intervention the had recieved - follow up would be done at 2, 6, and 12 week intervals.

Patients would be asked to fill 3 standardized questionnaires (translated to Hebrew and verified): PHQ-9, OHIP-14, ERQ . The clinical appearance of their lichen planus would be documented using a standardized semi-quantitive method as described by Piboonniyom et al, OOOO 2005

DETAILED DESCRIPTION:
Background:

Lichen planus (LP) is an immune-mediated skin and mucous membrane disease that mainly affects middle-aged adults of both sexes with a slight tendency to women. The precise prevalence of LP is unknown, but it is estimated that the oral form (OLP) alone is expressed in about 1-2% of the population. OLP is a chronic disease and it is considered by the World Health Organization (WHO) as a pre-malignant condition. OLP presents in five clinical forms - reticular, plaque-like, erythematous/atrophic, erosive/ulcerative and bullous. The reticular form is the most common and is characterized by white papules and/or white mesh-like stripes called Wickham's striae, typically bilaterally and symmetrically distributed. The most affected site is the posterior buccal mucosa followed by the tongue, gingiva and labial mucosa.2 Usually, this condition is asymptomatic even if it is diffuse, but the erythematous, erosive and ulcerative forms might cause a painful burning sensation. In 1978 the WHO published diagnostic criteria for OLP based on clinical and histopathological characteristics and in 2003 van der Meij and van der Waal modified these criteria, which are accepted till this day.

Despite a vast number of studies, the etiology of OLP remains unknown. It is believed that OLP is a result of a local cell-mediated immune response, involving antigen-presenting cells and inflammatory infiltrate predominantly of T lymphocytes, but its precipitating factors have not been determined. Some conditions have been associated with OLP, including among others, genetic predisposition, specific microorganisms, several systemic health conditions, and emotional disorders. The latter have been thoroughly investigated and some studies have showed that OLP patients, especially those with the erythematous/erosive forms, have higher state of anxiety and depression than non-OLP individuals. It has been suggested that psychological factors can alter the functionality of the immune system, leading to the development of autoimmune diseases. To date, no study has conclusively demonstrated a cause-and-effect relationship and more investigations about the possible correlation of anxiety and emotions with the severity of OLP are needed.

Hypnosis is a natural human phenomenon and every human tends to have trance like events several times a day. Techniques for induction and deepening of the hypnotic trance can be utilized in order to maintain this state and access aspects of psyche and physiology that are not readily accessible in the ordinary waking state.

Ample literature is available on the use of hypnosis for treatment of medical conditions that are exacerbated by emotions such as autoimmune and autoinflammatory conditions. That being said there are only anecdotal reports of hypnotherapy being used for Lichen Planus of the skin and non for OLP.

Study design:

Patients with a histologically confirmed diagnosis of OLP for at least 1 year prior to participation and examined by Dr. Zlotogorski (AZ) or Dr. Whitefield (SW) would be offered to participate and would give signed consent.

Willing patients' presentation and behavior of OLP would be documented in a Clinical Research File (CRF) and clinically photographed. CRF would include frequency of need for topical/systemic steroids, retinoids, calcineurin inhibitors and a semiquantitive scoring system for monitoring oral lichenoid lesions (from Piboonniyom et al, OOOO 2005).

Questionnaires would be filled out.

All Patients would be given Hebrew versions standardized and validated questionnaires:

Emotion Regulation Questionnaire (ERQ), Patient Health Questionnaire (PHQ-9), Oral Health Impact Profile (OHIP-14).

At this point patients would be referred to Dr. Wasserman (GW) who is an oral medicine specialist and licensed to practice medical hypnosis as well as for research related to hypnosis by the hypnosis advisory committee to the ministry of health.

GW would conduct a test of hypnotisability using a pendulum and "magnetic fingers".

Patients who rank with low hypnotisability would be added to the control group.

Patients who rank well would be randomized into 2 groups:

1. Psychoeducation group
2. Psychoeducation and hypnosis group Randomization would be done by flipping a coin.

GW would administer a brief presentation of psychoeducation and the relevance of the psycho-neuro-immuno-endocrine system to OLP. Patients randomized for hypnosis would also receive an explanation about hypnosis. This is to establish rapport between GW and each patient. All patients would be instructed not to mention the contents of the session with GW to AZ or to SW.

For patients selected for hypnosis, a short interview would be conducted about themselves including hobbies, favorite practices and places, fears or dislikes, daily stressors and triggers, effect of OLP on their lives - this is to tailor metaphors and suggestions for each participant and to strengthen rapport.

Hypnosis would include:

* Induction.
* Hypnotic relaxation and escalating deepening of hypnotic trance.
* Suggestions for healing and wellness of the oral mucosa and for balanced and optimal performance of the immune system, tailoring metaphors and images based on interview with patients.

"…the interior of the mouth is soft, healthy pink, intact and whole. It functions optimally as it should - enabling joyful eating and tasting, speaking with ease for any needed expression, any function of the mouth that needs to be used can be done so easily.

The immune system is very wise - it knows perfectly how to function in a balanced and harmonious way. Its wisdom enables it to act if the body needs defense and to standby and rest if it does not".

* Ego strengthening.
* Anchoring - using a predetermined mark selected by the patient.
* Dehypnotisation.

After dehypnotisation patients would be guided through rapid trance induction by themselves using the anchor created while in trance.

In case of an abreaction during trance, patients would be excluded from the trial and referred to a psychologist.

At the end of the session patients would be instructed to practice self-hypnosis at least once a day and set a reminder on their phone. Patients selected for hypnosis would receive a weekly phone call to "nudge" the daily practice and also to record that number of times they practiced. The session would be documented under an "Oral Medicine - Research" admission and under "Research - confidential" on the hospital's electronic medical record platform.

Two weeks, 6 weeks, and 3 months after the session with GW, patients would be clinically reassessed by AZ or SW. They would receive a phone call or a text message as reminder not to mention the contents of their session with GW in order to secure the blinding.

On a day of follow up, questionnaires would be filled out, and AZ or SW would conduct a thorough clinical examination, enter data into the CRF and conduct photographic documentation.

As control 30 age matched OLP patients who meet the inclusion criteria but were not offered to participate or even told of the study would be analyzed retrospectively according to the medical record - all patients in the Oral Mucosal clinic would be documented using the same semiquantitive scoring system and NRS.

Data collected from these patients would include demographic information as well as their semiquantitive score which is always recorded for OLP patients. Data would be accessed from the "Chameleon" platform.

The data will be retrospectively collected and anonymously stored using a connecting list between the research code and the participants' details. Each participant will be given a number and the data will be typed into an electronic spreadsheet after all the identifying details have been deleted.

The connecting list will be kept in a locked closet of the PI, or in a password-protected computer at the hospital. The list will be destroyed once the data processing is complete. A note regarding that will be made at the report regarding the end of the research.

The separation of the identifying data will be made only by the PI or sub-PI, who is from the hospital's staff, with authorization to access medical files.

The file will not be sent by a non-encrypted e-mail and will be taken out of the hospital without signing a contract with the R&D division.

The data will be stored in an anonymous file for a period of 7 years after the termination of the study. The file will be password-protedcted on the departmental server.

Data analysis Data will be analyzed using SPSS 28 (IBM). T-test would be used for continuous variables, ANOVA test would be used to test variability between groups, Chi square for nominal variables and correlation tests between groups.

Statistical significance is defined as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically and clinically confirmed diagnosis of OLP.
* At least 1 year since diagnosis.
* Above 18 years of age.
* Fluent in Hebrew or English (for the purpose of hypnosis).
* Lesions that are consistent with OLP are clinically visible in oral cavity.

Exclusion Criteria:

* Under aged.
* Previous negative experience with hypnosis.
* Psychiatric diagnosis of schizophrenia, personality disorder, severe depression, or history of psychosis.
* Substantial cognitive decline.
* Low hypnotisability.
* Previous oral squamous cell carcinoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-29 (Estimated); Primary Completion 2026-11-29 (Estimated); Study Completion 2026-11-29 (Estimated)

PRIMARY OUTCOMES:
Improvement in clinical expression of Oral Lichen Planus | 3 months
  The investigators expect to see an improvement in the clinical manifestation of oral lichen planus in the hypnotherapy group by assessing the score of the semiquantitive scale as described by Piboonniyom et al OOOO 2005
Improvement in clinical expression of Oral Lichen Planus | 3 months
  The investigators expect to see an improvement in pain or discomfort of oral lichen planus in the hypnotherapy group as stated on a 0-10 Numerical Rating Scale (NRS).
Improvement in clinical expression of Oral Lichen Planus | 3 months
  The investigators expect to see an improvement in the overall experience of living with oral lichen planus in the hypnotherapy group as measured buy the OHIP-14 questionnaire.

SECONDARY OUTCOMES:
Stress reduction and overall improvement in quality of life | 3 months
  As assessed by questionnaires the investigators expect to see an improvement in stress and anxiety measured by the ERQ questionnaire.
Stress reduction and overall improvement in quality of life | 3 months
  As assessed by questionnaires the investigators expect to see an improvement in stress and anxiety measured by the PHQ-9 questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Oral Medicine Unit, Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Yes
Patients IDs would be masked. Demographics, questionnaires, semiquantitive lichen planus assesment score would be recoreded - all in a spreadsheet. Would be available upon request to a specific journal reviewer or scientist.
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Piboonniyom SO, Treister N, Pitiphat W, Woo SB. Scoring system for monitoring oral lichenoid lesions: a preliminary study. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2005 Jun;99(6):696-703. doi: 10.1016/j.tripleo.2004.07.013. PMID 15897856
- [Background] Shenefelt PD. Hypnosis in dermatology. Arch Dermatol. 2000 Mar;136(3):393-9. doi: 10.1001/archderm.136.3.393. PMID 10724204
- [Background] Day M, Clarke SA, Castillo-Eito L, Rowe R. Psychoeducation for Children with Chronic Conditions: A Systematic Review and Meta-analysis. J Pediatr Psychol. 2020 May 1;45(4):386-398. doi: 10.1093/jpepsy/jsaa015. PMID 32219409
- [Background] Marshall GD Jr, Agarwal SK, Lloyd C, Cohen L, Henninger EM, Morris GJ. Cytokine dysregulation associated with exam stress in healthy medical students. Brain Behav Immun. 1998 Dec;12(4):297-307. doi: 10.1006/brbi.1998.0537. PMID 10080859
- [Background] Zucoloto ML, Shibakura MEW, Pavanin JV, Garcia FT, da Silva Santos PS, Maciel AP, de Barros Gallo C, Souza NV, Innocentini LMAR, Humberto JSM, Motta ACF. Severity of oral lichen planus and oral lichenoid lesions is associated with anxiety. Clin Oral Investig. 2019 Dec;23(12):4441-4448. doi: 10.1007/s00784-019-02892-2. Epub 2019 Apr 15. PMID 30989337
- [Background] Vallejo MJ, Huerta G, Cerero R, Seoane JM. Anxiety and depression as risk factors for oral lichen planus. Dermatology. 2001;203(4):303-7. doi: 10.1159/000051777. PMID 11752817
- [Background] Alves MG, do Carmo Carvalho BF, Balducci I, Cabral LA, Nicodemo D, Almeida JD. Emotional assessment of patients with oral lichen planus. Int J Dermatol. 2015 Jan;54(1):29-32. doi: 10.1111/ijd.12052. Epub 2014 Sep 10. PMID 25209436
- [Background] Chaudhary S. Psychosocial stressors in oral lichen planus. Aust Dent J. 2004 Dec;49(4):192-5. doi: 10.1111/j.1834-7819.2004.tb00072.x. PMID 15762340
- [Background] Soto Araya M, Rojas Alcayaga G, Esguep A. Association between psychological disorders and the presence of Oral lichen planus, Burning mouth syndrome and Recurrent aphthous stomatitis. Med Oral. 2004 Jan-Feb;9(1):1-7. English, Spanish. PMID 14704611
- [Background] Rojo-Moreno JL, Bagan JV, Rojo-Moreno J, Donat JS, Milian MA, Jimenez Y. Psychologic factors and oral lichen planus. A psychometric evaluation of 100 cases. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 1998 Dec;86(6):687-91. doi: 10.1016/s1079-2104(98)90205-0. PMID 9868726
- [Background] McCartan BE. Psychological factors associated with oral lichen planus. J Oral Pathol Med. 1995 Jul;24(6):273-5. doi: 10.1111/j.1600-0714.1995.tb01181.x. PMID 7562664
- [Background] Kramer IR, Lucas RB, Pindborg JJ, Sobin LH. Definition of leukoplakia and related lesions: an aid to studies on oral precancer. Oral Surg Oral Med Oral Pathol. 1978 Oct;46(4):518-39. No abstract available. PMID 280847
- [Background] Warnakulasuriya S, Kujan O, Aguirre-Urizar JM, Bagan JV, Gonzalez-Moles MA, Kerr AR, Lodi G, Mello FW, Monteiro L, Ogden GR, Sloan P, Johnson NW. Oral potentially malignant disorders: A consensus report from an international seminar on nomenclature and classification, convened by the WHO Collaborating Centre for Oral Cancer. Oral Dis. 2021 Nov;27(8):1862-1880. doi: 10.1111/odi.13704. Epub 2020 Nov 26. PMID 33128420
- [Background] van der Meij EH, van der Waal I. Lack of clinicopathologic correlation in the diagnosis of oral lichen planus based on the presently available diagnostic criteria and suggestions for modifications. J Oral Pathol Med. 2003 Oct;32(9):507-12. doi: 10.1034/j.1600-0714.2003.00125.x. PMID 12969224